CLINICAL TRIAL: NCT00663403
Title: Pharmacokinetics of Daptomycin in Critically Ill Patients Receiving Continuous Venovenous Hemodialysis (CVVHD)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Cubist Pharmaceuticals LLC, a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Responsible Party: Bruce A. Mueller, University of Michigan, College of Pharmacy
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: 063940; HUM00005646 (Other: U Michigan IRBMED)
Record Dates: First submitted 2008-04-18; First posted 2008-04-22 (Estimated); Results first posted 2010-08-26 (Estimated); Last update posted 2015-12-30 (Estimated); Status verified 2009-05

CONDITIONS: Critically Ill; Hemodialysis
Keywords: daptomycin; pharmacokinetics; renal replacement therapy; critical illness; intensive care units
MeSH Terms: conditions — Critical Illness | interventions — Daptomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Daptomycin — Daptomcyin 8 mg/kg infused intravenously every 48 hours
  Other Names: Cubicin

SUMMARY:
Daptomycin is an antibiotic that is affective against many strains of antibiotic resistant microorganisms. This antibiotic would be appropriate for use in the intensive care unit (ICU) considering the severity of illness and high risk for infection within this hospital environment. While in the ICU, patients may develop acute renal failure. Approximately 75% of ICU patients who develop acute renal failure will require some form of renal replacement therapy until their kidneys recover. Continuous hemodialysis is becoming one of the most common forms of dialysis in the ICU as it is a gentle type of dialysis provided over longer periods of time. The current data demonstrating the ability of continuous hemodialysis to remove daptomycin from the body is derived from in-vitro trials. The purpose of this trial is to determine the extent of daptomycin removal from critically ill patients receiving continuous hemodialysis. Findings from this trial will be used to develop new dosing recommendations for daptomycin in continuous hemodialysis.

DETAILED DESCRIPTION:
Daptomycin is a FDA approved antibiotic. This pharmacokinetic trial will monitor daptomycin drug concentrations during continuous hemodialysis. The daptomycin concentration profiles developed from this study will assist in developing a dose recommendation that will result in daptomycin levels that are safe and within therapeutic ranges, as previously identified, in critically ill patients with acute renal failure treated with continuous hemodialysis.

ELIGIBILITY:
Inclusion Criteria:

* =/> 18 years of age
* Prescribed Continuous Venovenous Hemodialysis (CVVHD) as determined by the primary physician
* Prescribed daptomycin as determined by the primary physician
* Informed consent granted

Exclusion Criteria:

* < 18 years of age
* Allergy to daptomycin
* Patients being primarily treated with daptomycin for diagnosis of osteomyelitis, meningitis, or pneumonia without adequate concomitant use of other more effective antimicrobial agents as daptomycin is not indicated for primary treatment of these types of infections
* Inability to complete 48 hours of Continuous Venovenous Hemodialysis (CVVHD)
* Concurrent use of other extracorporeal therapies such as Extracorporeal Membrane Oxygenation (ECMO) or plasmapheresis and intermittent hemodialysis
* Inability to obtain informed consent
* Pregnant and/or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2007-02; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruce A Mueller, PharmD, Principal Investigator — University of Michigan, College of Pharmacy
Locations (1):
- University of Michigan University Hospital, Ann Arbor, Michigan, United States

REFERENCES:
- [Derived] Vilay AM, Grio M, Depestel DD, Sowinski KM, Gao L, Heung M, Salama NN, Mueller BA. Daptomycin pharmacokinetics in critically ill patients receiving continuous venovenous hemodialysis. Crit Care Med. 2011 Jan;39(1):19-25. doi: 10.1097/CCM.0b013e3181fa36fb. PMID 20890189

RESULTS

PARTICIPANT FLOW:
Groups:
- Daptomycin in Continuous Renal Replacement Therapy (CRRT): This is a single arm study. Critically ill study subjects receiving continuous venovenous hemodialysis and prescribed daptomycin will receive daptomycin 8 mg/kg IV every 48 hours. Serial serum and effluent samples will be collected over 48 hours to assess daptomycin transmembrane clearance and pharmacokinetics during continuous venovenous hemodialysis.
Period: Overall Study
Arm/Group | Daptomycin in Continuous Renal Replacement Therapy (CRRT)
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Daptomycin in Continuous Renal Replacement Therapy (CRRT)
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 51 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 5
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Daptomycin Transmembrane Clearance by Continuous Venovenous Hemodialysis
Description: Quantifies the rate of daptomcyin removal by continuous venovenous hemodialysis.
Time Frame: From time of daptomycin administration to 48 hours post dose when subjects were also receiving continuous venovenous hemodialysis
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | Daptomycin in Continuous Renal Replacement Therapy (CRRT)
Number analyzed (Participants) | 8
mL/min | 6.3 (2.9)

2. Secondary Outcome: Daptomycin Dose Actually Administered
Time Frame: Time of daptomycin administration
Measure: Mean (Standard Deviation); unit: mg/kg
Arm/Group | Daptomycin in Continuous Renal Replacement Therapy (CRRT)
Number analyzed (Participants) | 8
mg/kg | 7.7 (0.6)

3. Secondary Outcome: Observed Daptomycin Peak Serum Concentration
Description: The maximum concentration of daptomycin in the body after receiving a dose of the drug. This was determined at the end of the daptomycin intravenous infusion at approximately 30 min.
Time Frame: At the end of the daptomycin intravenous infusion (at approximately 30 minutes)
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Daptomycin in Continuous Renal Replacement Therapy (CRRT)
Number analyzed (Participants) | 8
ug/mL | 81.2 (19.0)

4. Secondary Outcome: Daptomycin Volume of Distribution at Steady State
Description: Volume of distribution quantifies the distribution of daptomycin between the blood and the rest of the body. The greater the volume of distribtion, the greater the extent of daptomycin distribution throughout the body.
Time Frame: From time of daptomycin administration to 48 hours post dose
Measure: Mean (Standard Deviation); unit: L/kg
Arm/Group | Daptomycin in Continuous Renal Replacement Therapy (CRRT)
Number analyzed (Participants) | 8
L/kg | 0.23 (0.14)

5. Secondary Outcome: Daptomycin Total Body Clearance
Description: Total body clearance represents the rate at which daptomycin is removed from the body. In patients treated with continuous venovenous hemodialysis, the major pathways of daptomycin removal likely are: removal by continuuous venovenous hemodialysis (transmembrane clearance) and breakdown by the liver.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: mL/min/kg
Arm/Group | Daptomycin in Continuous Renal Replacement Therapy (CRRT)
Number analyzed (Participants) | 8
mL/min/kg | 0.13 (0.04)

6. Secondary Outcome: Daptomycin Half-life
Description: Half-life describes the time it takes for the concentration of the daptomycin in the body to decrease by one half.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Daptomycin in Continuous Renal Replacement Therapy (CRRT)
Number analyzed (Participants) | 8
hours | 20.8 (16.5)

7. Secondary Outcome: Daptomycin Free Fraction
Description: In the body, daptomcyin may be bound to proteins in the blood or it may not be bound to any proteins (also as the "free" component.) Free fraction describes the percent of daptomycin that is unbound or free. The unbound portion of daptomycin is able to kill bacteria.
Time Frame: From time of daptomycin administration to 48 hours post dose
Measure: Mean (Standard Deviation); unit: percent protein binding
Arm/Group | Daptomycin in Continuous Renal Replacement Therapy (CRRT)
Number analyzed (Participants) | 8
percent protein binding | 17.5 (5.0)

ADVERSE EVENTS:
Time Frame: From time of daptomycin administration to 48 hours post dose
Arm/Group | Daptomycin in Continuous Renal Replacement Therapy (CRRT)
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 0/8

LIMITATIONS AND CAVEATS:
Transmembrane and total body clearance results limited to continuous venovenous hemodialysis run at ~2 L/h dialysate flow. Clinical outcomes (such as infection cure rate, length of hospital stay, mortality rate) of subjects was not assessed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No